CLINICAL TRIAL: NCT04424615
Title: Idiopathic Granulomatous Mastitis
Acronym: IGM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif M Bakeer, head of general surgery department, Assiut University
Other Study IDs: IGM
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Granulomatous Mastitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of incidence, diagnosis and treatment of idiopathic granulomatous mastitis in Assiut university hospital

DETAILED DESCRIPTION:
Idiopathic granulomatous mastitis is an uncommon, benign and chronic inflammatory breast disease that mainly involves women of childbearing age . The disease, was first described by Kessler and Wollock in 1972 .Although it is a benign condition, it is important from different points of view: it poses a diagnostic and treatment dilemma , also, it clinically and mammographically mimics breast cancer, especially inflammatory type . On the other hand, due to lack of a definitive treatment plan, complications of empiric treatment, such as allergic reaction to antibiotics and poor cosmetic procedures result in following repeated surgical interventions which threaten the patients . In fact, the etiology of IGM is unknown but some factors have been stated including reaction to chemical materials such as oral contraceptive pills, infectious disease, autoimmune diseases and immunologic response formilk leakage from the breast's lobule . On the other hand, some conditions such as pregnancy, breast feeding, hyper prolactinemia, galactorrhea, and alpha 1 antitrypsin deficiency have been associated with the risk of the disease . Infection with corynebacterium kroppenstedtii has been suggested but is unconfirmed . The final word about etiology is that although the cause of the disease is unknown the general consensus is that reproductive age, recent pregnancy, breast feeding and history of oral contraceptive pills use are the most associated conditions with the disease, as shown in finding. The most common presenting sign is a defined hard lump of the breast. As the disease progresses nipple inversion, peau d'orange, tumorous in duration, ulcer and fistula can occur that can easily be mistaken for cancer . The most common reported ultrasound (U/S) findings are: an irregular hypo echoic finding that connects with the tubular hypo echo area and parenchymal heterogeneity and an area of mixed echo pattern with parenchymal deformity, both of which can lead to diagnosis of malignant changes . Common findings in mammography imaging are asymmetric diffuse and skin thickness . As mentioned previously, neither U/S nor mammography can differentiate IGM from malignant or other benign lesions, especially inflammatory breast cancers . Because of U/S and mammographic failure, some authors suggested MRI in diagnosis of IGM, but studies have shown that MRI does not provide additional findings for differentiation of IGM from breast cancer. In view of the non-definitive clinical and imaging findings, histopathology is the cornerstone of definitive diagnosis . It must be mentioned that FNA cannot confidently differentiate IGM and histopathological examination remains as the cornerstone . Some studies obtained different results in terms of the treatment of these patients that suggested corticosteroids and methotrexate with surgery or treatment with corticosteroid and azithromycin, and administration of steroids in lesions in these patients .

ELIGIBILITY:
Inclusion Criteria:

1- patients proved idiopathic granulomatous mastitis by histopathological examinaton 2 - Patients during child bearing period

Exclusion Criteria:

1. - tuberculous mastitis, ductectasi, fat necrosis, fungal infection, and sarcoidosis were excluded.
2. - post-surgical granulomatous reactions against foreign material

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients during child bearing period
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
clinical response rate | six months
  The clinical response is categorized into ''completely healed,'' ''inadequately healed,'' ''stable,'' ''worsened,'' or ''relapsed'' if the lesions had once healed but symptoms returned.
  clinical response rate [ Time Frame: six months ] The clinical response is categorized into ''completely healed,'' ''inadequately healed,'' ''stable,'' ''worsened,'' or ''relapsed'' if the lesions had once healed but symptoms returned.

SECONDARY OUTCOMES:
recurrence rate | two years
  granulomatous mastitis recurrence

REFERENCES:
- [Background] Bellavia M, Damiano G, Palumbo VD, Spinelli G, Tomasello G, Marrazzo A, Ficarella S, Bruno A, Sammartano A, Fiorentini T, Scio A, Maione C, Lo Monte AI. Granulomatous Mastitis during Chronic Antidepressant Therapy: Is It Possible a Conservative Therapeutic Approach? J Breast Cancer. 2012 Sep;15(3):371-2. doi: 10.4048/jbc.2012.15.3.371. Epub 2012 Sep 28. PMID 23091553
- [Background] Garcia-Rodiguez JA, Pattullo A. Idiopathic granulomatous mastitis: a mimicking disease in a pregnant woman: a case report. BMC Res Notes. 2013 Mar 14;6:95. doi: 10.1186/1756-0500-6-95. PMID 23497626
- [Background] Kalayci TO, Koruyucu MB, Apaydin M, Etit D, Varer M. Idiopathic Granulomatous Mastitis Associated with Erythema Nodosum. Balkan Med J. 2016 Mar;33(2):228-31. doi: 10.5152/balkanmedj.2015.150089. Epub 2016 Mar 1. PMID 27403395